CLINICAL TRIAL: NCT00505622
Title: A Multi-centre, Open Label Extension Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Perampanel (E2007) as an Adjunctive Therapy in Levodopa Treated Parkinson's Disease Subjects With Motor Fluctuations
Brief Title: Evaluation of the Long-term Safety, Tolerability, and Efficacy of Perampanel (E2007) as an Adjunctive Therapy in Levodopa Treated Parkinson's Disease Subjects With Motor Fluctuations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-318; 2007-000801-30 (EudraCT Number)
Record Dates: First submitted 2007-07-09; First posted 2007-07-23 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

ARMS (1):
- E2007 (Experimental): E2007 2 mg (one 2 mg tablet taken daily in the evening), or 4 mg (two 2 mg tablets daily in the evening).
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel

SUMMARY:
This is a multicentre, open-label extension study to evaluate the long-term safety, tolerability, and efficacy of Perampanel (E2007) as an adjunctive therapy in levodopa treated PD subjects with motor fluctuations. All subjects who have completed E2007-E044-213 or E2007-G000-309 will be candidates for entering this extension trial, provided that they meet the inclusion/exclusion criteria and have completed the core study, up to and including the final efficacy visit.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female subjects with idiopathic PD who have fulfilled the entry criteria to studies E2007-G000-309 or E2007-E044-213.

Subjects must have completed the core efficacy study up to and including the final efficacy and follow up visits as applicable.

Subjects with mild or moderate AEs thought to be related to Perampanel (E2007) can be entered into the study if the investigator considers it safe.

EXCLUSION CRITERIA:

1. Show evidence of clinically significant disease (i.e., severe cardiovascular or pulmonary disease, bronchial asthma, endocrine disease, history of peptic ulcer disease, history of myocardial infarction with residual atrial nodal or ventricular arrhythmias) that, in the opinion of the investigator, could affect either the patient's safety or the conduct of the study.
2. Pregnant or lactating women.
3. Women of childbearing potential (WOCBP) unless infertile (including surgically sterile) or practicing effective contraception (e.g., intrauterine device [IUD] or barrier method plus hormonal method). These subjects must have a negative urine pregnancy test at Visit 1 or 2 as indicated by entry into the study. These subjects must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non-child bearing potential as determined by the investigator.
4. Subjects with a past (within the past 5 years) or present history of drug or alcohol abuse as per Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM IV) criteria.
5. Antipsychotics are permitted as necessary. Subjects may be taking anti-depressant medication, however the dose must be stable for 4 weeks prior to their first study visit (the visit at which the inclusion and exclusion criteria are done with the patient).
6. Subjects with a past (within one year) or present history of major depression, suicidal ideation, or suicide attempts.
7. Subjects with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastrointestinal, haematological, endocrine, or metabolic systems that might complicate assessment of the tolerability of the study medication.
8. Subjects with significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper limit of the normal range).
9. Subjects with current or prior treatment (within 4 weeks prior to the Screening Visit) with medication known to induce the enzyme CYP3A4.
10. Clinically significant ECG abnormality, and/or prolonged QTc (defined as QTc ≥ 450 msec).
11. Current or prior treatment (within 4 weeks prior to entry visit) with tolcapone, methyldopa, budipine, or reserpine.
12. Subjects with previous stereotactic surgery (e.g., pallidotomy) for PD or with planned stereotactic surgery during the study period
13. Subjects receiving or with planned (next 12 months) deep brain stimulation.
14. Subjects with conditions affecting the peripheral or central sensory system unless related to PD (such as mild sensory or pain syndromes limited to OFF periods) that could interfere with the evaluation of any such symptoms caused by the study medication.
15. Subjects have received an investigational product (other than E2007 or entacapone 200 mg) within 4 weeks prior to Screening
16. Any condition that could, in the opinion of the investigator, place the subject at increased risk or is likely to prevent completion of the study.
17. Subjects with any condition that would make the subject, in the opinion of the investigator, unsuitable for the study.
18. Patients on pergolide or cabergoline.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, MD, Study Director — Eisai Inc.
Locations (1):
- Centre d'Investigation Clinique, Hospital Purpan, Toulouse, Toulouse Cedex, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel (Placebo During Core Study); Perampanel (Entacapone 200mg During Core Study); Perampanel (Perampanel 4mg During Core Study): Subjects entered this open-label extension study from the double-blind core study (E2007-G000-309). Subjects started on perampanel 2mg once daily for 2 weeks, followed by 4mg once daily for 2 weeks (Titration Phase); Subjects then continued onto the maintenance phase of perampanel 4mg once daily for 2 weeks. Subjects who did not tolerate the study drug at 4mg were allowed to down-titrate to 2mg. Subjects who did not tolerate 2mg were withdrawn from the study.
Period: Overall Study
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Started | 121 | 108 | 96
Completed | 0 | 0 | 0
Not Completed | 121 | 108 | 96
Not completed — Adverse Event | 5 | 6 | 4
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Study termination by sponsor | 115 | 98 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study) | Total
Number analyzed (Participants) | 121 | 108 | 96 | 325
Age, Customized [Number; unit: Particpants] — Data comes from previous double-blind core study (E2007-G000-309). Safety Population.
  Particpants
    <65 | 65 | 52 | 46 | 163
    >= 65 | 56 | 56 | 50 | 162
Sex: Female, Male [Count of Participants; unit: Participants] — Data comes from previous double-blind core study (E2007-G000-309). Safety Population - All subjects entering the open-label extension study who took at least 1 dose of perampanel.
  Participants
    Female | 46 | 44 | 30 | 120
    Male | 75 | 64 | 66 | 205
Race/Ethnicity, Customized [Number; unit: participants] — This baseline characteristic is for Race. Data comes from previous double-blind core study (E2007-G000-309). Safety Population.
  participants
    White | 92 | 75 | 65 | 232
    Asian | 29 | 33 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Daily OFF Time (Hours) During Open-label Extension Study
Description: OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor. All data was collected using a 3-day diary within a window of a defined visit.
Time Frame: Baseline, Week 0, Week 2, Week 4, Week 8, Week 20, Follow-up
Population: Safety Population - All subjects entering the open-label extension study who took at least 1 dose of perampanel.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Number analyzed (Participants) | 121 | 108 | 96
Hours
  Week 0 | -1.03 (2.635) | -1.07 (2.595) | -1.24 (2.643)
  Week 2 | -0.91 (2.323) | -1.28 (2.867) | -1.31 (2.779)
  Week 4 | -0.65 (2.945) | -1.15 (2.010) | -1.67 (2.438)
  Week 8 | -0.70 (2.983) | -1.16 (2.509) | -1.36 (2.324)
  Week 20 | -1.34 (2.972) | -1.14 (1.805) | -2.11 (2.163)
  Follow-up | -0.77 (2.983) | -1.61 (2.435) | -0.94 (2.978)

2. Secondary Outcome: Mean Change From Baseline in UPDRS Part II (ADL) Score in OFF State (Hours) During Open-label Extension Study
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part II assesses activities of daily living (ADL) based on 13 items, such as speech, hygiene, and falling. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 0, Week 20, Week 32
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Number analyzed (Participants) | 121 | 108 | 96
Scores on a scale
  Week 0 | -0.84 (4.241) | -1.99 (4.469) | -1.66 (4.598)
  Week 20 | -0.12 (4.727) | -2.82 (4.086) | -2.66 (4.972)
  Week 32 | 1.11 (2.667) | 0.60 (2.408) | -0.67 (3.141)

3. Secondary Outcome: Mean Change From Baseline in UPDRS Part III (Motor) Score in ON State (Hours) During Open-label Extension Study
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. ON state is when medication is providing benefits to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 0, Week 20, Week 32
Population: Safety population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Number analyzed (Participants) | 121 | 108 | 96
Scores on a scale
  Week 0 | -0.25 (6.874) | -0.64 (6.911) | -0.96 (6.999)
  Week 20 | 0.30 (7.463) | -0.53 (6.950) | -1.63 (8.005)
  Week 32 | 2.22 (5.869) | -2.00 (5.523) | 7.17 (6.463)

4. Secondary Outcome: Mean Change From Baseline in Total Daily ON Time (Without Dyskinesias or With Non-troublesome Dyskinesias) (Hours) During Open-label Extension Study
Description: ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor. All data was collected using a 3-day diary within a window of a defined visit.
Time Frame: Baseline, Week 0, Week 2, Week 4, Week 8, Week 20, Follow-up
Population: Safety population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Number analyzed (Participants) | 121 | 108 | 96
Hours
  Week 0 | 1.08 (2.820) | 0.58 (3.004) | 0.48 (2.773)
  Week 2 | 0.30 (2.776) | 0.80 (2.731) | 0.91 (2.940)
  Week 4 | 0.38 (2.825) | 0.43 (2.091) | 1.24 (2.724)
  Week 8 | 0.17 (3.099) | 0.52 (2.542) | 0.73 (2.261)
  Week 20 | 0.94 (3.535) | 0.82 (2.231) | 1.62 (2.351)
  Follow-up | 0.43 (3.368) | 1.12 (2.561) | 0.85 (3.497)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were defined as treatment emergent in this study if the start date of the event was on or after the start of study medication in this study. Adverse events that occurred 30 days after the last dose of study drug were 'post-treatment'.
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Entacapone 200mg During Core Study) | Perampanel (Perampanel 4mg During Core Study)
Serious Adverse Events (participants affected / at risk) | 2/121 | 6/108 | 2/96
Other Adverse Events (participants affected / at risk) | 27/121 | 27/108 | 17/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=121) | Perampanel (Entacapone 200mg During Core Study) (N=108) | Perampanel (Perampanel 4mg During Core Study) (N=96)
Dementia (Nervous system disorders) | 0 | 1 | 0
Parkinson's Disease (Nervous system disorders) | 1 | 0 | 0
Radicular Syndrome (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=121) | Perampanel (Entacapone 200mg During Core Study) (N=108) | Perampanel (Perampanel 4mg During Core Study) (N=96)
Dizziness (Nervous system disorders) | 8 | 3 | 4
Dyskinesia (Nervous system disorders) | 4 | 6 | 5
On and Off Phenomenon (Nervous system disorders) | 9 | 12 | 6
Parkinson's Disease (Nervous system disorders) | 7 | 3 | 1
Somnolence (Nervous system disorders) | 4 | 6 | 3

LIMITATIONS AND CAVEATS:
Due to early termination, no subjects completed this open-label extension study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No